CLINICAL TRIAL: NCT04074226
Title: Erector Spinae Plane (ESP) Block With Liposomal Bupivacaine Versus Quadratus Lumborum (QL) Block With Liposomal Bupivacaine for Postoperative Pain Management After Open Total Abdominal Hysterectomy: A Prospective Randomized Controlled Trial
Brief Title: ESP vs QL for Total Abdominal Hysterectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Inability to recruit patients for the past several months due to all the staffing shortages and changes to the surgeons' practice patterns
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, John Alexander, Associate Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: STU-2019-1174
Record Dates: First submitted 2019-07-26; First posted 2019-08-30 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Postoperative Pain
Keywords: regional anesthesia; postoperative pain; erector spinae plane block; quadratus lumborum block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: No other parties will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ultrasound-guided ESP block with liposomal bupivacaine (Experimental): For the ESP block, the transducer will be placed parasagittally at the level of the tip of the scapula and the anesthesiologist will scan in a craniocaudal manner to identify the ipsilateral T10 transverse process and overlying erector spinae muscle. Following aseptic preparation of the injection site and the ultrasound probe, a 22-gauge, 10mm block needle will be introduced parallel to the ultrasound guided beam (in-plane technique) until its tip reaches the plane between the erector spinae muscle and transverse process. After negative aspiration, 20 ml of a mixture containing 10ml 0.25% bupivacaine and 10ml 1.3% liposomal bupivacaine will be injected in 5 ml increments to separate the fascial plane between the muscle and transverse process. The investigators will observe local anesthetic spread under real-time imaging. The block will then be performed in the same manner on the opposite site.
  Interventions: Procedure: Erector Spinae Plane block
- Ultrasound-guided QL block with liposomal bupivacaine (Active Comparator): For the QL block, the transducer will be placed transversely over the lumbar spine at the level of the iliac crest. Then, the anesthesiologist will scan laterally to identify the ipsilateral L3 transverse process, psoas muscle, and quadratus lumborum muscle to identify the "Shamrock Sign" (7). Following aseptic preparation of the injection site and the ultrasound probe, a 22-gauge, 10mm block needle will be introduced parallel to the ultrasound guided beam (in-plane technique) until its tip reaches the plane between the quadratus lumborum muscle and psoas muscle. After negative aspiration, 20 ml of a mixture containing 10ml 0.25% bupivacaine and 10ml 1.3% liposomal bupivacaine will be injected in 5 ml increments to separate the fascial plane between the two muscles. The investigators will observe local anesthetic spread under real-time imaging. The block will then be performed in the same manner on the opposite site.
  Interventions: Procedure: Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Erector Spinae Plane block — The Erector Spinae Plane (ESP) block is a new block first described in 2016 which blocks terminal branches of the lower thoracic and lumbar nerve roots. It is performed by injection of local anesthetic in the fascial plane below the erector spinae muscle group.
  Arms: Ultrasound-guided ESP block with liposomal bupivacaine
Procedure: Quadratus Lumborum Block — Ultrasound-guided QL block has been reported to provide effective analgesia in patients undergoing lower abdominal surgical procedures, including in patients undergoing abdominal hysterectomy. Ultrasound guidance offers a number of advantages, including the ability to visualize the anatomy, perform real-time navigation, and direct observation of local anesthetic spread. The QL block is performed via ultrasound-guided injection of local anesthetic in the fascial planes above or below the QL muscle
  Arms: Ultrasound-guided QL block with liposomal bupivacaine

SUMMARY:
Patients undergoing open total abdominal hysterectomy (n=82) at Parkland Memorial Hospital will be randomized into one of two groups to receive either ultrasound-guided bilateral ESP block with liposomal bupivacaine (Group 1) or ultrasound-guided bilateral QL block with liposomal bupivacaine (Group 2) for postoperative pain management. The remaining aspect of perioperative care, including the general anesthetic technique and postoperative care will be standardized and will be similar for all patients. The duration of the involvement in the study will be until 72 hours postoperatively. Anesthesia providers will identify potential subjects during their Pre-Anesthesia Evaluation Clinic visit and/or Day Surgery Unit pre-anesthetic assessment. There will be no incentive or payment to the patients.

Patients in Group 1 will receive ultrasound-guided bilateral ESP block in the preoperative holding area prior to surgery. Patients in Group 2 will receive ultrasound-guided QL block in the preoperative holding area prior to surgery. All patients will have general anesthesia per previously established Parkland Enhanced Recovery After Surgery (ERAS) protocols. Postoperatively, patients in both Groups will receive acetaminophen 1000 mg orally every 8 hours, meloxicam 15 mg orally every 24 hours, and immediate-release oxycodone 5 - 10mg orally every 4 hours as needed for breakthrough pain.

The postoperative analgesia will be documented using the Numeric Rating Scale (0-10 scale where 0=no pain and 10=worst pain). In addition, total opioid dose over the 72-hours study period will be documented. Postoperative nausea will be measured using a categorical scoring system (none=0, mild=1, moderate=2, severe=3) and episodes of vomiting will be documented. Rescue anti-emetics will be given to any patient who complains of nausea and/or vomiting. All variables will be assessed at 4, 6, 12, 24, 48, and 72 hours, postoperatively by an investigator blinded to group allocation.

DETAILED DESCRIPTION:
The investigators will study 82 American Society of Anesthesiologists (ASA) physical status 1-3 subjects scheduled for open Total Abdominal Hysterectomy who will be identified by anesthesia providers during their Pre-Anesthesia Evaluation Clinic visit and/or Day Surgery Unit pre-anesthetic assessment at Parkland Hospital. If the subjects agree to participate in the study, the researchers will determine eligibility. If the subject meets all inclusion/exclusion criteria, the subject will be asked to sign the Consent Form and HIPAA Authorization Form prior to any study procedures in a face-to-face meeting with the researchers.

Protected patient information will include name, medical record number, date of birth, and contact information including telephone number. Height and weight will also be recorded. All patients will receive a standardized general anesthetic based on Enhanced Recovery After Surgery protocols. One of the investigators will randomly allocate patients using computer generated randomization schedule to one of the two groups.

Study Groups:

Group 1: Ultrasound-guided ESP block with liposomal bupivacaine

Group 2: Ultrasound-guided QL block with liposomal bupivacaine.

Anesthesiologists with previous experience in ultrasound-guided regional anesthesia procedures will perform the block based on randomization results. In both groups the patient will be placed in a sitting position, a SonoSite X-Porte linear ultrasound transducer will be used for real-time ultrasound guidance.

Group 1: For the QL block, the transducer will be placed transversely over the lumbar spine at the level of the iliac crest. Then, the anesthesiologist will scan laterally to identify the ipsilateral L3 transverse process, psoas muscle, and quadratus lumborum muscle to identify the "Shamrock Sign" (7). Following aseptic preparation of the injection site and the ultrasound probe, a 22-gauge, 10mm block needle will be introduced parallel to the ultrasound guided beam (in-plane technique) until its tip reaches the plane between the quadratus lumborum muscle and psoas muscle. After negative aspiration, 20 ml of a mixture containing 10ml 0.25% bupivacaine and 10ml 1.3% liposomal bupivacaine will be injected in 5 ml increments to separate the fascial plane between the two muscles. The investigators will observe local anesthetic spread under real-time imaging. The block will then be performed in the same manner on the opposite site.

Group 2: For the ESP block, the transducer will be placed parasagittally at the level of the tip of the scapula and the anesthesiologist will scan in a craniocaudal manner to identify the ipsilateral T10 transverse process and overlying erector spinae muscle. Following aseptic preparation of the injection site and the ultrasound probe, a 22-gauge, 10mm block needle will be introduced parallel to the ultrasound guided beam (in-plane technique) until its tip reaches the plane between the erector spinae muscle and transverse process. After negative aspiration, 20 ml of a mixture containing 10ml 0.25% bupivacaine and 10ml 1.3% liposomal bupivacaine will be injected in 5 ml increments to separate the fascial plane between the muscle and transverse process. The investigators will observe local anesthetic spread under real-time imaging. The block will then be performed in the same manner on the opposite site.

A standard postoperative analgesic regimen in both groups will include acetaminophen 1000 mg, orally every 8 hours and meloxicam 15mg, orally every 24 hours. For breakthrough pain (or rescue), immediate-release oxycodone 5-10mg, orally every 4 hours as needed for pain will be provided.

The efficacy of postoperative analgesia will be documented in all patients using the visual analog score (0=no pain, 10=worst pain). In addition, total morphine dose over the 72-hours study period will be documented. Postoperative nausea will be measured using a categorical scoring system (none=0, mild=1, moderate=2, severe=3) and episodes of vomiting will be documented. Rescue antiemetics will be given to any patient who complains of nausea or vomiting. All variables will be assessed at 4, 6, 12, 24, 48, and 72 hours postoperatively by an investigator blinded to group allocation.

For each patient the following data will be recorded:

Preoperatively:

* Age
* Gender
* Height
* Weight
* Baseline pain score
* Pre-operative block procedure, duration, amount of analgesia used
* Time to perform the blocks

Intraoperatively:

• Surgical time

Postoperatively:

* Post-Anesthesia Care Unit time
* Post-operative pain scores at 4, 6, 12, 24, 48, 72 hours
* cumulative opioid consumption during the first 24-hours postoperatively
* Time to first ambulation
* Time to first oral intake
* Time to be ready for discharge home

ELIGIBILITY:
Inclusion Criteria:

* Female ASA physical status 1-3 scheduled for open abdominal hysterectomy
* Age 18-80 years old
* Able to participate personally or by legal representative in informed consent in English or Spanish

Exclusion Criteria:

* History of relevant drug allergy
* Age less than 18 or greater than 80 years
* Chronic opioid use or drug abuse
* Active use of anticoagulant medication
* Significant psychiatric disturbance
* Inability to understand the study protocol
* Refusal to provide written consent

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Study population is for hysterectomy (surgical removal of the uterus) which is only present in female patients
Enrollment: 17 (Actual)
Dates: Start 2021-03-20 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-03-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain (NRS = numeric rating scale) at 24 hours | 24 hours
  The primary aim of this study is to compare postoperative pain scores at 24 hours between the subjects who receive ESP block with liposomal bupivacaine and the subjects who receive QL block with liposomal bupivacaine undergoing Total Abdominal Hysterectomy. The investigators will use the Numeric Rating Scale, measuring patient report of pain from 0 = no pain up to 10 = worst possible pain.

SECONDARY OUTCOMES:
Postoperative Pain (NRS = numeric rating scale) at 48 hours | 48 hours
  One secondary objectives is to compare pain scores at 48 hours. The investigators will use the Numeric Rating Scale, measuring patient report of pain from 0 = no pain up to 10 = worst possible pain.
Postoperative Pain (NRS = numeric rating scale) at 72 hours | 72 hours
  Another secondary objective is to compare pain scores at 48 hours and 72 hours. The investigators will use the Numeric Rating Scale, measuring patient report of pain from 0 = no pain up to 10 = worst possible pain.
Opioid Use (oral morphine equivalents) | 24 hours
  Another secondary objective is to assess cumulative opioid consumption during the first 24-hours postoperatively. The investigators will convert all opioids consumed in this time from to oral morphine equivalents.
Block Time (minutes) | 1 hour
  Antoher secondary objective is to assess the time to perform the blocks as measured in minutes.
Ambulation Time (hours:minutes) | 24 hours
  Another secondary objective is to assess the time to first ambulation as measured in hours:minutes after the end of surgery.
Oral Intake Time (hours:minutes) | 24 hours
  Another secondary objective is to assess the time to first oral intake as measured in hours:minutes after the end of surgery.
Discharge Readiness Time (hours:minutes) | 72 hours
  Another secondary objective is to assess the time time for discharge readiness as measured in hours:minutes after the end of surgery.

CONTACTS AND LOCATIONS:
Overall Officials: John C Alexander, MD, Principal Investigator — UT Southwestern
Locations (1):
- Parkland Health and Hospital System, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data will not be shared

REFERENCES:
- [Background] Elsharkawy H, Bajracharya GR, El-Boghdadly K, Drake RL, Mariano ER. Comparing two posterior quadratus lumborum block approaches with low thoracic erector spinae plane block: an anatomic study. Reg Anesth Pain Med. 2019 Mar 28:rapm-2018-100147. doi: 10.1136/rapm-2018-100147. Online ahead of print. PMID 30923253
- [Background] Elsharkawy H, El-Boghdadly K, Barrington M. Quadratus Lumborum Block: Anatomical Concepts, Mechanisms, and Techniques. Anesthesiology. 2019 Feb;130(2):322-335. doi: 10.1097/ALN.0000000000002524. No abstract available. PMID 30688787
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016